CLINICAL TRIAL: NCT04768283
Title: Evaluation of Cardiac Rehabilitation Functional and Physical Capacity, Health-related Quality of Life and Associations With Frailty in Older Patients After Ischemic Heart Disease and Interventional Treatment
Brief Title: Cardiac Rehabilitation and Additional Physical Training in Elderly Patients After Acute Coronary Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Aurelija Beigienė, Aurelija Beigienė, MD, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-12-19 BE-2-107
Record Dates: First submitted 2021-02-21; First posted 2021-02-24 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Frailty Syndrome; Ischaemic Heart Disease
Keywords: Frailty; Cardiac surgery; Cardiac rehabilitation; Exercise training; Resistance training; Balance training
MeSH Terms: conditions — Frailty; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Cardiac rehabilitation physical training program included: respiratory muscle training (7 days/week, for 15 minutes) and aerobic exercises on cycle ergometers (6 days/week, for 10-30 minutes, 30-50% watts or 30-50% HRmax).
- Intervention group 1 (Experimental): Combinated physical training program:
  Respiratory exercises, aerobic training will be the same as in the control group.
  Additional exercises: balance training and strength exercises with weights, elastic resistance rubbers.
  Interventions: Other: Additional balance and resistance training - 1
- Intervention group 2 (Experimental): Combinated physical training program:
  Respiratory exercises, aerobic training will be the same as in the control group.
  Additional exercises: balance training with static and dynamic balance training device Biodex Balance System TM SD and strength exercises with HUR strength training machines.
  Interventions: Other: Additional balance and resistance training - 2

INTERVENTIONS:
Other: Additional balance and resistance training - 1 — Additional exercise program with balance and resistance training three times per week.
  The balance training included exercises to improve static as well as dynamic balance ability, for 15-20 minutes.
  The resistance training included exercises with weights (0,5, 1 or 2 kg), elastic resistance rubbers, intensity 30-50% 1-RM, 10 repetitions with 3 sets and 3 minute rest between sets.
  Arms: Intervention group 1
Other: Additional balance and resistance training - 2 — Additional exercise program with balance and resistance training three times per week.
  The balance training included exercises with static and dynamic balance training device Biodex Balance System TM SD, for 15-20 minutes. Exercises are performed with the following programs: Postural stability training, Limits of stability training, Weight shift training, Maze control training, Random control training, Percent weight-bearing training.
  The resistance training included exercises with HUR strength training machines, intensity 30-50% 1-RM, 10 repetitions with 3 sets and 3 minute rest between sets. Strength training was performed with the following exercises: Leg press, leg extension, leg abduction, leg adduction.
  Arms: Intervention group 2

SUMMARY:
The aim of this study is to evaluate functional and physical capacity, health-related quality of life and associations with frailty in older patients after ischemic heart disease and interventional treatment with an individualized physical training program in the second phase of cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients after acute coronary syndrome and percutaneous coronary intervention or coronary bypass surgery;
* Age 65 years and older;
* 6-minute walk distance (6-MWD) ≥150 meters;
* Left ventricular ejection fraction ≥ 40%;
* Patient's agreement to participate in the study.

Exclusion Criteria:

* combined coronary artery bypass grafting and valve surgery;
* Cardiac devices;
* Diseases in the musculoskeletal system or other organs complicating physical activity and exercise training;
* Exercise-limiting comorbidities (primarily orthopedic and neurological conditions that would exclude individuals from participating in cardiac rehabilitation according to study protocol), cognitive or linguistic deficits.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Frailty level by Edmonton frail scale score | baseline
  Frailty measured by The Edmonton frail scale score - 0-3 - fit, 4-5 - vulnerable, 6-7 - mild frailty, 8-9 - moderate frailty,10-17 - severe frailty.
Change from baseline functional capacity by six minutes walking test (6MWT) | baseline, 3 weeks
  6MWT measured by meters
Change from baseline cardiopulmonary exercise capacity by maximal load (maxWatt) | baseline, 3 weeks
  Maximal load measured with spiroergometry by maximal watts
Change from baseline cardiopulmonary exercise capacity by maximal oxygen consumption (peakVO2) | baseline, 3 weeks
  PeakVO2 measured with spiroergometry by millilitres of oxygen per kilogram of body mass per minute
Change from baseline quality of life by MacNew questionnaire | baseline, 3 weeks
  The MacNew Heart Disease HRQL questionnaire consists of 27 items which fall into three domains (a 13-item physical limitations domain scale, a 14-item emotional function domain scale, and a 13-item social function domain scale). There are 5 items that inquire about symptoms: angina/chest pain, shortness of breath, fatigue, dizziness, and aching legs. The time frame for the MacNew is the previous two weeks.

SECONDARY OUTCOMES:
Change from baseline physical performance by Short Physical Performance Battery (SPPB) | baseline, 3 weeks
  The short physical performance battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests.The scores range from 0 (worst performance) to 12 (best performance).
Change from baseline muscular strength by one repetition maximum test (1RM) | baseline, 3 weeks
  1RM test for leg extension measured by kilograms

CONTACTS AND LOCATIONS:
Locations (1):
- LUHS hospital Kaunas Clinics Rehabilitation hospital of Kulautuva, Kulautuva, Kaunas County, Lithuania

IPD SHARING:
Plan to Share IPD: No